CLINICAL TRIAL: NCT07017725
Title: A Dose-escalation and Safety Study of CID-103 Followed by a Randomized, Open-label, Parallel-arm Multi-dose Study Evaluating the Efficacy and Tolerability of CID-103 in Adults With Chronic Immune Thrombocytopenia
Brief Title: A Dose-escalation Study Followed by a Dose Optimal Study to Evaluate the Safety and Efficacy of CID-103 in Adults With Chronic Immune Thrombocytopenia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CASI-CID-103-201; CTR20244168 (Registry Identifier: Chinese Clinical Trial Register (ChiCTR))
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Chronic Immune Thrombocytopenia
Keywords: Purpura; Thrombocytopenic; Idiopathic
MeSH Terms: conditions — Purpura

STUDY DESIGN:
Intervention Model Description: Part A (Dose Escalation and Safety Phase): This phase combines the accelerated escalation and traditional 3+3 escalation with at least five dosing cohorts designed:30 mg, 150 mg, 300 mg, 600 mg, and 900 mg. Subjects will receive an initial priming dose of either 30 mg for the first two cohorts or 150 mg for the rest of cohorts. Dose escalation to the next cohort will be determined based on safety and tolerability data.
  Part B (Randomized Dose Comparison Phase): This phase follows a parallel assignment model, in which participants are randomly assigned to one of three selected doses of CID-103: low, intermediate, or high. The purpose is to determine the optimal dose to advance into future studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part B (Randomized Dose Exploration) high-dose cohort (Experimental): Each participant will receive selected high-dose. Once approximately 8 evaluable subjects per arm have completed approximately six weeks of treatment, an initial review of safety and efficacy will be conducted by the SMC to determine if there is one or more sub-optimal dose(s) that should be closed to further recruitment or if dose / regimens require adjustment.
  Interventions: Drug: CID-103
- Part B (Randomized Dose Exploration) intermediate-dose cohort (Experimental): Each participant will receive selected intermediate-dose. Once approximately 8 evaluable subjects per arm have completed approximately six weeks of treatment, an initial review of safety and efficacy will be conducted by the SMC to determine if there is one or more sub-optimal dose(s) that should be closed to further recruitment or if dose / regimens require adjustment.
  Interventions: Drug: CID-103
- Part B (Randomized Dose Exploration) low-dose cohort (Experimental): Each participant will receive selected low-dose. Once approximately 8 evaluable subjects per arm have completed approximately six weeks of treatment, an initial review of safety and efficacy will be conducted by the SMC to determine if there is one or more sub-optimal dose(s) that should be closed to further recruitment or if dose / regimens require adjustment.
  Interventions: Drug: CID-103
- Part A (Dose Escalation) Cohort 1- 30 mg/30 mg (Experimental): This is the initial dose cohort with accelerated dose escalation design. If a Grade ≥ 2 AE is reported in the cohort, the cohort will expand to three subjects and the study will then convert to a standard 3+3 design.
  Interventions: Drug: CID-103
- Part A (Dose Escalation) Cohort 1- 30 mg/150 mg (Experimental): This is the second dose cohort with accelerated dose escalation design. If a Grade ≥ 2 AE is reported in the cohort, the cohort will expand to three subjects and the study will then convert to a standard 3+3 design.
  Interventions: Drug: CID-103
- Part A (Dose Escalation) Cohort 1- 150 mg/300 mg (Experimental): This is the third dose cohort with accelerated dose escalation design. If a Grade ≥ 2 AE is reported in the cohort, the cohort will expand to three subjects and the study will then convert to a standard 3+3 design.
  Interventions: Drug: CID-103
- Part A (Dose Escalation) Cohort 1- 150 mg/600 mg (Experimental): This is the fourth dose cohort with standard 3+3 design.
  Interventions: Drug: CID-103
- Part A (Dose Escalation) Cohort 1- 150 mg/900 mg (Experimental): This is the fifth dose cohort with standard 3+3 design.
  Interventions: Drug: CID-103

INTERVENTIONS:
Drug: CID-103 — Strength:20 mg/mL. Route of administration: IV infusion. Treatment duration: QW for 6 weeks, then at the same dose Q2W up to Week 12. If treatment continues after Week 12, dosing will occur monthly for up to a maximum treatment duration of six months.

SUMMARY:
The goal of the global Phase 1/2 clinical trial is to evaluate whether CID-103, a novel anti-CD38 monoclonal antibody, is safe and effective in adults with chronic immune thrombocytopenia (ITP). The main questions the study aims to answer are:

* To evaluate the safety and tolerability of CID-103 in subjects with ITP with different increasing doses of CID-103.
* To further evaluate the safety and tolerability of CID-103 at two or three dose levels and to select an optimal dose and administration regimen for CID-103 for further study of clinical efficacy.

The study will be done in two parts:

Part A will test increasing doses of CID-103 to see how safe it is and how well people tolerate it. Researchers will also aim to find a safe dose range.

Part B will compare up to three different doses of CID-103 to see how well the medicine works and gather more safety and efficacy information. The goal is to find the optimal dose to use in future studies.

CID-103 is given through an intravenous (IV) infusion. During the study, participants may receive treatment for up to 6 months, followed by a post-treatment safety follow-up period to check for ongoing safety and effectiveness.

This study is an important step toward developing a new treatment for people living with chronic ITP. If CID-103 is found to be safe and effective, it could offer a new option for patients who do not respond well to current therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female individuals aged 18 to 65 years at time of signing of ICF. Disease-related.
2. Diagnosed with ITP that has persisted for ≥ 3 months, diagnosed in accordance with The American Society of Hematology 2019 Guidelines for Immune Thrombocytopenia or the Updated International Consensus Report on the Investigation and Management of Primary Immune Thrombocytopenia (as locally applicable).
3. Diagnosis of ITP supported by a prior response to an ITP treatment (other than a thrombopoietin receptor agonists [TPO-RA]) that achieved a platelet count of ≥ 30 x 10^9/L and a doubling of baseline measurement.
4. Has received at least two lines of SOC systemic treatment (i.e., corticosteroids and one other agent).
5. Has a mean platelet count ≤ 35 x 10^9/L on at least two measurements at least one week apart during screening.
6. If receiving standard background treatment for ITP, treatment should be stable in dose and frequency for at least four weeks prior to first dose of CID-103.
7. Adequate organ function.
8. Contraception: Female participants must either be non-pregnant or not breastfeeding and must have a negative pregnancy test. Male and female participants must meet the contraceptive requirements.

Exclusion Criteria:

1. Prior treatment with any anti-CD38 agent, or has been treated with anti-Bruton's tyrosine kinase (BTK), neonatal Fc receptor (FcRn) antagonist or complement inhibitor within three months prior to first dose of CID-103.
2. Use of IV immunoglobulin, subcutaneous immunoglobulin or anti-D immunoglobulin treatment within four weeks of screening.
3. Treatment with rituximab or splenectomy within the three months prior to first dose of CID-103.
4. Use of anticoagulants or any drug with antiplatelet effect (such as aspirin) within three weeks before screening.
5. Receiving other concurrent investigational therapies or have received investigational therapies within four weeks of the first dose of CID-103 or five half-lives (if shorter).
6. Active hemolytic anemia.
7. Diagnosed with severe chronic obstructive pulmonary disease (COPD), Global Initiative for Chronic Obstructive Lung Disease (GOLD Stage 3 or 4) or asthma.
8. Has been diagnosed with myelodysplastic syndrome or other active malignancy.
9. Known / clinically significant amyloidosis.
10. Has a history of any thrombotic or embolic event within six months before screening.
11. A history or evidence of cardiovascular risk including left ventricular ejection fraction < 50%, clinically significant uncontrolled ventricular arrhythmia, acute coronary syndrome history, coronary angioplasty or stenting within six months, current ≥ Class III congestive heart failure (NYHA guidelines), and treatment refractory hypertension.
12. Clinically significant medical history or ongoing chronic illness.
13. Known active infection with hepatitis B (HBV) (surface antigen) or infection with hepatitis C (HCV) in absence of sustained virologic response.
14. History of known or suspected immunosuppression.
15. Known active infection with human immunodeficiency virus (HIV) and CD4+ T cell count < 350/μL.
16. Karnofsky Performance Status ≤ 70.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of CID-103 | 10 months
  * Occurrence of DLTs (Part A only)
  * Frequency of TEAEs
  * Related AEs
  * Grade 3/4 AEs
  * Serious adverse events (SAEs)
  * Fatal AEs
  * AEs leading to CID-103 discontinuation up to Week 12
  * Percentage of subjects with at least one treatment-related Grade ≥ 3 TEAE, SAE or AE leading to CID-103 discontinuation up to Week 12 (Part B only)
Platelet response | 12 weeks
  A platelet count ≥ 50 x 10^9/L and ≥ 20 x 10^9/L above baseline achieved on at least two consecutive measurements at least seven days apart.

SECONDARY OUTCOMES:
Platelet count | 12 weeks
  The secondary efficacy endpoint is Platelet count, defined as platelet count ≥ 30 x 10^9/L and > 2-fold increase in platelet count from baseline and absence of bleeding requiring medical intervention / treatment, measured on at least two consecutive occasions at least seven days apart.
Complete platelet response | 12 weeks
  The secondary efficacy endpoint includes percentage of subjects with complete platelet response, defined as platelet count ≥ 100 x 109/L and absence of bleeding requiring medical intervention / treatment, measured on at least two consecutive occasions at least seven days apart.

CONTACTS AND LOCATIONS:
Overall Officials: Junping Chen, Study Chair — CASI pharmaceutical, Inc
Locations (6):
- China (6):
  - North China University of Science and Technology Affiliated Hospital, Tangshan, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan